CLINICAL TRIAL: NCT02865174
Title: Comparison of Topical Tranexamic Acid and Floseal® on Blood Loss After Total Knee Arthroplasty in Patients With a Thromboembolic Risk
Brief Title: Topical Tranexamic Acid and Floseal® in Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wang Jun-Wen, Wang Jun-Wen [wang0155], Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NMMRPG8F0191
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Thrombin-gelatin matrix; Floseal; Tranexamic Acid; Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Tranexamic Acid; Tranylcypromine; FloSeal Matrix; Enoxaparin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Topical tranexamic acid (Active Comparator): Intraarticular application of tranexamic acid Enoxaparin for venous thromboembolism prophylaxis in the duration of hospital stay
  Interventions: Drug: Topical tranexamic acid; Drug: Enoxaparin
- Floseal® (Active Comparator): Floseal® was applied on potential bleeding sites before prosthesis implantation.
  Enoxaparin for venous thromboembolism prophylaxis in the duration of hospital stay
  Interventions: Drug: Floseal®; Drug: Enoxaparin
- Control group (Placebo Comparator): No intervention before closure of joint capsule. Enoxaparin for venous thromboembolism prophylaxis in the duration of hospital stay
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Topical tranexamic acid — Intraarticular application of tranexamic acid 3g in 100 ml normal saline into knee joint after closure of the joint capsule
  Other Names: Topical transamine
  Arms: Topical tranexamic acid
Drug: Floseal® — Floseal® (Hemostatic matrix, 10ml, Baxter) was applied on potential bleeding sites: the femoral insertion of the posterior cruciate ligament, the lateral genicular artery after resection of the meniscus, the posterior capsule of the knee joint, the bony surfaces not covered by the implant as well as the pinholes (femur and tibia). The entire content of a 10 mL vial containing the active product (Floseal®) was used. The HM remained in place for 3 minutes and was then gently rinsed from the knee as recommended by the manufacturer (Baxter)
  Other Names: Thrombin-gelatin matrix
  Arms: Floseal®
Drug: Enoxaparin — Enoxaparin will be administrated sc 40mg each day postoperatively as venous thromboembolism prophylaxis in the duration of hospital stay
  Other Names: Low molecular weight heparin

SUMMARY:
Our purpose of this study is to conduct a prospective randomized controlled trial to investigate the blood-conservation effect of this two topical hemostatic agents in primary TKA procedures in patients with a risk of thromboembolic events. We will also observe if there is increased risk of thromboembolism by use of topical hemostatic agents.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is associated with considerable blood loss and increasing needs for allogenic blood transfusion. Previous studies demonstrated a transfusion rates ranging from 10% to 38% after standard TKAs. Transfusion carries significant risks of cardiopulmonary embarrassment, disease transmission, immunological reaction and postoperative infection.

The major causes of postoperative blood loss following TKA are attributed to surgery itself which induces a considerable activation of the coagulation cascade and local fibrinolysis, the latter is further enhanced after release of the tourniquet at the end of surgery. Tranexamic acid (TXA), an inhibitor of fibrinolysis, was reportedly effective reducing blood loss after standard TKA. Our previous experiences in minimally invasive (MIS) TKA showed that intraoperative infusion of TXA reduced 45% of postoperative blood loss and needs for transfusion from 20% to 4%. However, most of the orthopedic surgeons still hesitate to use TXA systemically in TKAs especially in high risk patients with a potential increase in thromboembolic events following surgery. A recent study by Nishihara et al demonstrated that use of TXA in total hip arthroplasty did not appear to affect the prevalence of either proximal DVT or PE. Another study by Xie J et al also showed the incidence of postoperative VTE was unchanged when TXA was administered in primary unilateral TKA, but in there study the total occurrence of vascular occlusive events was statistically significantly higher (17.55% Vs 9.35%, p < 0.001) in the TXA group. However, in this two studies the patient with high risk of thromboembolic events (ischemic heart disease, chronic renal failure on hemodialysis, cerebral infarction, previous VTE disease, thrombophilia associated with genetic diseases) were excluded.

We believe the topical use of hemostatic agent in patients with high risk of thromboembolism can avoid its systematic effect and decrease its potential perioperative risk of thromboembolic complications (arterial thrombosis, myocardial infarction and pulmonary embolism). Recently, there were some reports demonstrating the cost-effectiveness of topical application of TXA in TKA patients. Besides, thrombin-based hemostatic agents, Floseal®, have been widely used in surgical procedure including gynecology, general surgery, and orthopedics which were still attracting the attention and interest of multitudinous surgeons. Some recent studies demonstrated that topic use of Floseal® in primary TKA can reduce hemoglobin decline and calculated total blood loss after TKA and is not related to adverse reactions or complications such as wound infection, venous thromboembolism events(VTE). But there were another studies showed Floseal® does not reduce blood loss in TKA procedures.

Our purpose of this study therefore is to conduct a prospective randomized controlled trial to investigate the blood-conservation effect of this two topic hemostatic agents and their safety in a primary TKA procedures in patients with risk of thromboembolic events. The first group by topical TXA application, the second group by topical Floseal® application, and the third group of placebo and observe whether there is difference in the the blood-conservation effect by total blood loss calculation, hemoglobin loss and transfusion requirement among these patient groups.

ELIGIBILITY:
Inclusion Criteria:

History of ischemic heart disease, stroke, or VTE high risk group, such as obesity, varicose vein of the leg, previous history of PE or DVT, hypercoagulability, recent or ongoing treatment for cancer.

After cardiologist or neurologist's evaluation, patients who was classified as low-risk of perioperative risk Advanced knee osteoarthritis, Failure of medical treatment or rehabilitation. Hemoglobin > 11g/dl, No use of non-steroid anti-inflammatory agent one week before operation

Exclusion Criteria:

Preoperative Hemoglobin ≦11 g/dl History of infection or intraarticular fracture of the affective knee Renal function deficiency (GFR < 30 ml/min/1.73m2) Elevated liver enzyme, history of liver cirrhosis, impaired liver function and coagulopathy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Total blood loss after operation | From the operation to the postoperative day 3 or 4
  Total blood loss was calculated according to Nadler et al., which used maximum postoperative reduction of the Hb level adjust for weight and height of the patient. The formula is as follows, Total blood loss = (Total blood volume x [change in Hb level / preoperative Hb level])x1000+volume transfused
Decrease of hemoglobin level after operation | From the operation to the postoperative day 14
  We will check hemoglobin preoperatively and postop. Day 1, 2, 3 or 4 and 14. We will calculate the change of hemoglobin level on postoperative day 1, 2, 4, and 14.

SECONDARY OUTCOMES:
Incidence of major postoperative bleeding | within 30 days of the operation
  Major bleeding was defined as bleeding that involved a critical organ, or that required reoperation or clinically overt bleeding outside the surgical site that was associated with a decrease in the hemoglobin level of 2 g or more per deciliter or requiring infusion of 2 or more units of blood
Incidence of any non-major bleeding | within 30 days of the operation
  Non-major bleeding including hemorrhagic wound complications (excessive wound hematoma or bleeding at the surgical site
Incidence of wound infection after surgery | within 30 days of the operation
  composite of wound poor healing, superficial wound infection, and deep infection requiring return to surgery
Incidence of any thrombotic events | within 30 days of the operation
  the composite of any venous thromoembolism events, ischemic heart attacks, cerebrovascular accidents

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Wen Wang, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Koahsiung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gomez-Barrena E, Ortega-Andreu M, Padilla-Eguiluz NG, Perez-Chrzanowska H, Figueredo-Zalve R. Topical intra-articular compared with intravenous tranexamic acid to reduce blood loss in primary total knee replacement: a double-blind, randomized, controlled, noninferiority clinical trial. J Bone Joint Surg Am. 2014 Dec 3;96(23):1937-44. doi: 10.2106/JBJS.N.00060. PMID 25471907
- [Background] Schwab PE, Thienpont E. Use of a haemostatic matrix does not reduce blood loss in minimally invasive total knee arthroplasty. Blood Transfus. 2015 Jul;13(3):435-41. doi: 10.2450/2015.0199-14. Epub 2015 Jan 26. PMID 25761324
- [Background] Helito CP, Gobbi RG, Castrillon LM, Hinkel BB, Pecora JR, Camanho GL. Comparison of Floseal(r) and electrocautery in hemostasis after total knee arthroplasty. Acta Ortop Bras. 2013;21(6):320-2. doi: 10.1590/S1413-78522013000600004. PMID 24453689
- [Background] Comadoll JL, Comadoll S, Hutchcraft A, Krishnan S, Farrell K, Kreuwel HT, Bechter M. Comparison of hemostatic matrix and standard hemostasis in patients undergoing primary TKA. Orthopedics. 2012 Jun;35(6):e785-93. doi: 10.3928/01477447-20120525-14. PMID 22691647
- [Background] Kim HJ, Fraser MR, Kahn B, Lyman S, Figgie MP. The efficacy of a thrombin-based hemostatic agent in unilateral total knee arthroplasty: a randomized controlled trial. J Bone Joint Surg Am. 2012 Jul 3;94(13):1160-5. doi: 10.2106/JBJS.K.00531. PMID 22623075
- [Background] Suarez JC, Slotkin EM, Alvarez AM, Szubski CR, Barsoum WK, Patel PD. Prospective, randomized trial to evaluate efficacy of a thrombin-based hemostatic agent in total knee arthroplasty. J Arthroplasty. 2014 Oct;29(10):1950-5. doi: 10.1016/j.arth.2014.05.025. Epub 2014 Jun 5. PMID 25015756
- [Background] Di Francesco A, Flamini S, Fiori F, Mastri F. Hemostatic matrix effects on blood loss after total knee arthroplasty: A randomized controlled trial. Indian J Orthop. 2013 Sep;47(5):474-81. doi: 10.4103/0019-5413.118203. PMID 24133307
- [Background] Testini M, Marzaioli R, Lissidini G, Lippolis A, Logoluso F, Gurrado A, Lardo D, Poli E, Piccinni G. The effectiveness of FloSeal matrix hemostatic agent in thyroid surgery: a prospective, randomized, control study. Langenbecks Arch Surg. 2009 Sep;394(5):837-42. doi: 10.1007/s00423-009-0497-5. Epub 2009 May 7. PMID 19421770
- [Background] Clapp M, Huang JC. Use of FloSeal Sealant in the Surgical Management of Tubal Ectopic Pregnancy. Case Rep Obstet Gynecol. 2013;2013:906825. doi: 10.1155/2013/906825. Epub 2013 May 29. PMID 23819082
- [Background] Gazzeri R, Galarza M, Alfier A. Safety biocompatibility of gelatin hemostatic matrix (Floseal and Surgiflo) in neurosurgical procedures. Surg Technol Int. 2012 Dec;22:49-54. PMID 22915500
- [Background] Georgiadis AG, Muh SJ, Silverton CD, Weir RM, Laker MW. A prospective double-blind placebo controlled trial of topical tranexamic acid in total knee arthroplasty. J Arthroplasty. 2013 Sep;28(8 Suppl):78-82. doi: 10.1016/j.arth.2013.03.038. Epub 2013 Jul 29. PMID 23906869
- [Background] Konig G, Hamlin BR, Waters JH. Topical tranexamic acid reduces blood loss and transfusion rates in total hip and total knee arthroplasty. J Arthroplasty. 2013 Oct;28(9):1473-6. doi: 10.1016/j.arth.2013.06.011. Epub 2013 Jul 23. PMID 23886406
- [Background] Chimento GF, Huff T, Ochsner JL Jr, Meyer M, Brandner L, Babin S. An evaluation of the use of topical tranexamic acid in total knee arthroplasty. J Arthroplasty. 2013 Sep;28(8 Suppl):74-7. doi: 10.1016/j.arth.2013.06.037. PMID 24034510
- [Background] Wind TC, Barfield WR, Moskal JT. The effect of tranexamic acid on blood loss and transfusion rate in primary total knee arthroplasty. J Arthroplasty. 2013 Aug;28(7):1080-3. doi: 10.1016/j.arth.2012.11.016. Epub 2013 Mar 28. PMID 23541868
- [Derived] Yen SH, Lin PC, Wu CT, Wang JW. Comparison of Effects of a Thrombin-Based Hemostatic Agent and Topical Tranexamic Acid on Blood Loss in Patients with Preexisting Thromboembolic Risk Undergoing a Minimally Invasive Total Knee Arthroplasty. A Prospective Randomized Controlled Trial. Biomed Res Int. 2021 Jan 14;2021:2549521. doi: 10.1155/2021/2549521. eCollection 2021. PMID 33511201